CLINICAL TRIAL: NCT04214561
Title: Assessment of Sleep Structure, Selected Blood Parameters, Respiratory Function, Genotype, Phenotype, Pain, Anxiety and Psychosomatization in Patients With Bruxism
Brief Title: Relationship Between Selected Parameters and Bruxism
Acronym: WMU1/2019
Status: Enrolling by invitation | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Principal Investigator, Wroclaw Medical University
Other Study IDs: WMU1/2019
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Sleep Bruxism; Sleep Disorder; Psychosomatic Disorder; Pain; Anxiety; Mental Status Change; Temporomandibular Disorder
MeSH Terms: conditions — Sleep Bruxism; Sleep Wake Disorders; Psychophysiologic Disorders; Pain; Anxiety Disorders; Temporomandibular Joint Disorders | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SB group: Patients diagnosed with SB.
  Interventions: Diagnostic Test: Polysomnography
- Healthy controls: Patients without diagnosed SB.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Each of the patients will undergo polysomnography

SUMMARY:
Bruxism is a common phenomenon. It is estimated that its prevalence in the adult population is 8-31%. Bruxism occurring during sleep is the activity of the masticatory muscles that appear during sleep, which can be rhythmic or phased and is not a movement disorder or sleep disorder in healthy people. It is currently believed that bruxism should not be considered a disorder. In healthy people, it is treated rather as behavior, which may be a risk factor for pathological clinical implications or a protective factor in the presence of other disease entities. The most common symptoms of bruxism include: pathological wear and tooth sensitivity, periodontal and oral mucosa damage, myalgia in the stomatognathic system, headache and prosthetic restoration damage. However, due to nocturnal occurrence, bruxism symptoms may go unnoticed for a long time, which means that patients are often unaware of this behavior. The etiology of bruxism is multifactorial and not fully understood. It is currently believed that it can be caused by genetic, psychological and exogenous factors. Due to the unclear etiology of bruxism, it is so important to conduct research that allows making a certain diagnosis and finding the causes of this phenomenon

DETAILED DESCRIPTION:
Sleep breathing disorders are a frequent and serious health problem in the Polish population. Obstructive sleep apnea (OSA) is a common disorder. The essence of OSA is repeated episodes of airway obstruction that occur repeatedly during sleep, resulting in a decrease in the level of partial oxygen in the blood. Increased tension in the upper respiratory muscles and throat vibrations often result in very loud snoring. Apnea episodes end with awakenings that cause sleep fragmentation, deep sleep deficiency, and REM phase. Such episodes occur repeatedly, over a dozen or even several dozen times per hour of sleep. The consequence of episodes of obstruction and fragmentation of sleep is ineffective, restless sleep, pathological daytime sleepiness, falling asleep against your own will, awakening with a feeling of stopping breath, shortness of breath or choking. Sleep fragmentation and repetitive episodes of hypoxia result in poor quality of life, chronic fatigue and an increased risk of traffic accidents. The direct consequences of apnea are blood hypoxia, increased heart rate and increased blood pressure. Common complications of OSA are hypertension, stroke, arrhythmias, coronary artery disease, pulmonary hypertension and heart failure. Untreated OSA increases the risk of premature death, especially in men under 50 years of age, contributing to the development of vascular endothelial dysfunction and an increase in cardiovascular risk.

The causal relationship between bruxism and apnea has not been clearly established so far. There is also a lack of research on the contribution of genetic factors to the emergence and severity of both conditions.The project will be implemented at the Sleep Laboratory at the Clinic of Internal, Occupational Diseases and Hypertension of the Medical University of Wrocław, which has a technical room with three computer stations, three polysomnographic devices. About 100 patients will be examined at the Department of Internal Diseases, Occupational and Hypertension and Clinical Oncology because of suspected bruxism during sleep. The full polysomnographic examination with video recording will be directed to patients from the Chewing Organ Dysfunction Clinic operating at the Department of Experimental Dentistry at the Medical University of Wrocław, who will be interviewed and have a comprehensive external and intra-oral examination according to Diagnostic Criteria for Temporomandibular Disorders (DC / TMD) and based on the guidelines of the American Academy of Sleep Medicine International Classification of Sleep Disorders, probable bruxism during sleep will be diagnosed. Polysomnograms will be evaluated in 30-second folds, according to standard sleep criteria. PSG results will include data on sleep latency, total sleep time (TST) and sleep performance (%) as well as assessment of the N1, N2, N3 and REM phases. Respiratory pathological events will be assessed according to the American Sleep Academy standards. Apnea will be defined as no airflow through the airways for more than 10 seconds. Shortness of breath will be defined as a reduction in respiratory amplitude by more than 30% for more than 10 seconds, with subsequent blood desaturation by more than 3%, or with subsequent awakening. The activity of the masticatory muscles during the examination will be assessed on the basis of EMG recording from electrodes placed on the chin and symmetrically in the vicinity of the masseter muscles attachments. As episodes of bruxism, episodes of rhythmic activity of the masseter muscles, often accompanied by grinding or knocking noises and characteristic movements in the orofacial region occurring after a minimum interval of three seconds from the last muscular activity, will be qualified. Bruxism episodes will be assessed quantitatively using the BEI (Bruxism Episodes Index) rating the number of bruxism episodes per hour of patient's sleep, and qualitatively for phase, tonic and mixed episodes. The results will then be analyzed for the incidence of RMMA directly related to bruxism episodes and their relationship to sleep apnea episodes, changes in blood pressure and heart rhythm to determine time and cause-effect relationships.

In addition, we will carry out the following surveys: ISI Insomnia Severity Scale, KPS sense of stress questionnaire , TEC Traumatic Experience Checklist. , mini COPE stress management questionnaire, CECS Courtauld Emotional Control Scale, AIS Accteptance of Illness Scale ,BAI Beck Anxiety Index, Short Questionnaire for Measuring the Big Five IPIP-BFM-20, McGill Pain Questionnaire, GCSP Graded Chronic Pain Scale. , PHQ-9 Patient Health Questionnaire, Pittsburgh Sleep Quality Index PSQI, STOP-Bang Apnea Risk Questionnaire, Beck Depression Inventory, PSS-10 Perceived Stress Scale -10, HIT-6 Headache Impact Test,GAD-7 Generalized Anxiety Disorder ,MIDAS scale for assessing functioning disorders in migraine.

Each patient will also be subjected to genetic blood laboratory tests to determine the occurrence of specific genotypes and phenotypes occurring in patients with bruxism.

The tests will be carried out in accordance with the CONSORTated (CONsolidated Standards of Reporting Trials) guidelines for RCT (Randomized Controlled Trial). Expected effects:

1. Assessment of the incidence of bruxism during sleep in patients with breathing disorders during sleep
2. Determination of changes in sleep structure in patients with bruxism.
3. Assessment of possible genetic basis in patients with bruxism
4. Assessment of psychosomatization in patients with bruxism.
5. Assessment of the level of anxiety and pain felt in patients with bruxism.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed sleep bruxism
* age between 18 and 70

Exclusion Criteria:

* age under 18
* age over 70
* terminal general diseases
* severe mental disorders
* taking drugs that could falsify polysomnography
* confirmed alcoholism
* drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with probable sleep bruxism referred to the Department of Internal Medicine, Occupational Diseases and Hypertension and Clinical Oncology for polysomnography. Healthy controls.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between bruxism and sleep structure by polysomnography. | 15.10.2019 - 31.12.2020
  Polysomnograms will be evaluated in a 30-second contributions, according to standard sleep criteria. PSG results will contain data on the latency of sleep, total sleep time (TST), sleep efficiency (%) and an evaluation of phases N1, N2, N3 and REM.

SECONDARY OUTCOMES:
Relationship between bruxism and insomnia assessed by Insomnia Severity Scale. | 15.10.2019 - 31.12.2020
  Each participant will fill in Insomnia Severity Scale. Questionnaire contains 5 questions, scored from 0 to 4 depending on the severity of ailments. Minimal score is 0, maximal score is 20. A total point value of up to 10 is considered the norm, while a score above 14 points indicates clinically significant insomnia.
Relationship between bruxism and sense of stress assessed by Sense of stress questionnaire - KPS questionnaire measuring the structure of stress sensations. sense of stress questionnaire. | 15.10.2019 - 31.12.2020
  Each participant will fill in KPS sense of stress questionnaire. The questionnaire consists of 27 statements; the subject determines the extent to which the statement relates to him using a five-point scale. It allows you to calculate the overall score of generalized stress levels, as well as three results related to the following dimensions: emotional tension, external stress and intrapsychic stress. The questionnaire also contains the scale of lies.
Relationship between bruxism and trauma asessed by Traumatic Experience Checklist. | 15.10.2019 - 31.12.2020
  Each participant will fill in Traumatic Experience Checklist comprising 29 different traumatic experiences. It assesses 5 types of trauma and 4 types of problems: emotional neglect, emotional abuse, body threat, sexual harassment, and sexual abuse, serious family problems , death or loss of a family member, body harm, and war experiences. Scoring includes computing two indexes (overall index of number of traumas experienced resulting from the sum of all items, and the total area of traumatic presence which is the sum of the 5 traumatic experiences areas); and three trauma severity indexes (determined by the impact of trauma and age when it occurred, and assembled into emotional, physical, and sexual trauma). The severity of total trauma can range from 0 to 13 (neglect and emotional abuse, physical abuse, and sexual harassment or abuse) or from 0 to 24 (body threat, pain, and bizarre/strange punishment).
Relationship between bruxism and coping with stress assessed by mini COPE- inventory to measure stress management. | 15.10.2019 - 31.12.2020
  Each participant will fill in mini COPE. Questionnaire consists of 28 statements that make up 14 stress coping strategies.Some testing strategies were divided into four categories and corresponding strategies (inventory scales): active coping (including: active coping, planning, positive reevaluation), helplessness (including: taking psychoactive substances, cessation of actions, blaming self), seeking support (including: seeking emotional support, seeking instrumental support), avoidance behaviors (including dealing with something else, denying, discharging). three strategies create independent factors (turning to religion, acceptance, sense of humor). The range of results for each statement ranges from 0 to 3 points. The calculation of the results consists in adding to each other points for the answers regarding two theorems that make up the given scale, and then dividing by 2.
Relationship between bruxism and emotional controll assessed by Courtauld Emotional Control Scale. | 15.10.2019 - 31.12.2020
  Each participant will fill in Courtauld Emotional Control Scale that consists of three subscales, each of them containing seven statements regarding the way of showing anger, depression, and anxiety. The scale is used to measure subjective control of anger, anxiety, and depression in difficult situations and designed to examine adults (both healthy and ill). CECS is a tool of self-description. Summing up the scores of all three subscales, the overall score of emotion control is established. The examination aims at defining to what degree an individual is convinced subjectively of ability to control his/her reactions in the situation of experiencing given negative emotions. The overall indicator of emotion control is within the range of 21-84 points. The higher the score, the greater the suppression of negative emotions.
Relationship between bruxism and illness accteptance assessed by Accteptance of Illness Scale. | 15.10.2019 - 31.12.2020
  Each participant will fill in Accteptance of Illness Scale. The scale is used to measure the degree of acceptance of the disease. It contains eight statements describing the negative consequences of poor health. Each statement is scored from 1 to 5, where 1 means strongly agree and 5 strongly disagree. The scale has no standards. The obtained result is compared with the average result of one of eight clinical groups. The scale is used to measure the degree of disease acceptance. It can apply to any disease. The greater the acceptance of the disease, the better the adaptation and the less sense of mental discomfort.
Relationship between bruxism and anxiety assessed by Beck Anxiety Index. | 15.10.2019 - 31.12.2020
  Each participant will fill in Beck Anxiety Index. The total score is calculated by finding the sum of the 21 items. Total score for all 21 symptoms that can range between 0 and 63 points. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and; 26 - 63 as "Severe".
Relationship between bruxism and personality assessed by International Personality Item Pool-Big Five Markers-20. | 15.10.2019 - 31.12.2020
  Each participant will fill in IPIP-BFM 20. The questionnaire measures five traits (Extraversion, Agreeableness, Conscientiousness, Emotional Stability, Intellect), and consists of 20 items.
Relationship between bruxism and pain assessed by McGill questionnaire. | 15.10.2019 - 31.12.2020
  Each participant will fill in McGill questionnaire that is composed of 78 words. Respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain).
Relationship between bruxism and pain assessed by Graded Chronic Pain Scale. | 15.10.2019 - 31.12.2020
  Each participant will fill in Graded Chronic Pain Scale. Scoring Criteria for Grading Chronic Pain Severity: Characteristic Pain Intensity is a 0 to 100 score derived from Questions 1 through 3:Mean (Pain Right Now, Worst Pain, Average Pain) X 10. Disability Score is 0 to 100score derived from Questions 4 through 6:Mean (Daily Activities, Social Activities, Work Activities) X 10. Disability Points: Add the indicated points for Disability Days (Question 7)and for Disability Score. Classification: GRADE 0- No TMD pain in prior 6 months. GRADE I-Low Intensity Characteristic Pain Intensity<50, Low Disability<3 Disability Point. GRADE II -High Intensity Characteristic Pain Intensity >50, LowDisability<3 Disability Points. GRADE III- High Disability3 to 4 Disability Points, Moderately Limiting (Regardless of Characteristic Pain Intensity). GRADE IV- High Disability 5 to 6 Disability Points, Severely Limiting (Regardless of Characteristic Pain Intensity).
Relationship between bruxism and depression assessed by Patient Health Questionnaire - 9. | 15.10.2019 - 31.12.2020
  Each participant will fill in Patient Health Questionnaire - 9. PHQ-9 total score for the nine items ranges from 0 to 27.Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Relationship between bruxism and sleep quality assessed by Pittsburgh Sleep Quality Index - a self-report questionnaire that assesses sleep quality over a 1-month time interval. | 15.10.2019 - 31.12.2020
  Each participant will fill in Pittsburgh Sleep Quality Index. The measure consists of 19 individual items, creating 7 components that produce one global score ranging from 0 to 21, where lower scores mean better sleep quality.
Relationship between bruxism and apnea risk assessed by STOP-Bang. | 15.10.2019 - 31.12.2020
  Each participant will fill in STOP-Bang questionnaire. The total score ranges from 0 to 8. The lower the score is, the lower the risk of occurrence Obstructive Sleep Apnea (OSA).
Relationship between bruxism and depression assessed by Beck Depression Inventory. | 15.10.2019 - 31.12.2020
  Each participant will fill in Beck Depression Inventory. The questionnaire is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The minimum total score is 0, the maximum total score is 63. Enables scoring: 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression.
Relationship between bruxism and perceived stress assessed by Perceived Stress Scale - 10. | 15.10.2019 - 31.12.2020
  Each participant will fill in Perceived Stress Scale -10. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. It can range from 0 to 40. Scores ranging from 0-13 would be considered low stress,14-26 would be considered moderate stress, 27-40 would be considered high perceived stress.
Relationship between bruxism and headache assessed by Headache Impact Test - 6. | 15.10.2019 - 31.12.2020
  Each participant will fill in Headache Impact Test - 6 . These responses are summed to produce a total score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent.
Relationship between bruxism and anxiety assessed by Generalized Anxiety Disorder -7. | 15.10.2019 - 31.12.2020
  Each participant will fill in Generalized Anxiety Disorder -7 that consists of 7 items. Total score ranges 0-21 points. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Relationship between bruxism and headache impact assessed by Migraine Disability Assessment questionnaire. | 15.10.2019 - 31.12.2020
  Each participant will fill in Migraine Disability Assessment questionnaire. Scoring includes adding the total number of days from questions 1-5. Grading includes: grade I (little or no disability) 0-5 days, grade II (mild disability) 6-10 days, grade III (moderate disability) 11-20 days, grade IV (severe disability) more than 21 days.
Relationship between bruxism and genotype and fenotype assessed in blood test. | 15.10.2019 - 31.12.2020
  Each participant will undergo genetical blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Mieszko Wieckiewicz, DMD, PhD, Study Chair — Wroclaw Medical University; Helena Martynowicz, MD, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Orzeszek S, Martynowicz H, Smardz J, Wojakowska A, Bombala W, Jenca A Jr, Wieckiewicz M. Relationship between pain, quality of sleep, sleep bruxism and patients' personality among individuals with reported orofacial pain. Sci Rep. 2025 Jul 11;15(1):25009. doi: 10.1038/s41598-025-09978-w. PMID 40640286
- [Derived] Orzeszek S, Martynowicz H, Smardz J, Wojakowska A, Bombala W, Mazur G, Wieckiewicz M. Assessment of sleep quality in patients with orofacial pain and headache complaints: A polysomnographic study. Dent Med Probl. 2024 Jul-Aug;61(4):549-562. doi: 10.17219/dmp/177008. PMID 38832763
- [Derived] Wieckiewicz M, Martynowicz H, Lavigne G, Lobbezoo F, Kato T, Winocur E, Wezgowiec J, Danel D, Wojakowska A, Mazur G, Smardz J. An exploratory study on the association between serotonin and sleep breathing disorders. Sci Rep. 2023 Jul 21;13(1):11800. doi: 10.1038/s41598-023-38842-y. PMID 37479853